CLINICAL TRIAL: NCT05392985
Title: Chemotherapy Versus Endocrine Therapy in Metastatic Breast Cancer Patients With Heterogeneous Estrogen Receptor Expression
Brief Title: Detection and Analysis of MBC With Heterogeneous ER Expression
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-20
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FES+-: MBC patients with both FES positive(+) and negative(-) lesions.

SUMMARY:
To investigate the treatment pattern and efficacy of MBC patients with ER heterogeneity using a novel convenient way of 18F-fluoroestradiol positron emission tomography/computed tomography (18F-FES PET/CT).

ELIGIBILITY:
Inclusion Criteria:

* Patients received 18F-FES PET/CT in Fudan University Shanghai Cancer Center from 2017-2021.
* Patients had both FES positive (FES+) and negative (FES-) lesions in FES exam.
* Patients received further treatment.

Exclusion Criteria:

* Incomplete medical records.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival

SECONDARY OUTCOMES:
Adverse events | 6 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided